CLINICAL TRIAL: NCT01906060
Title: Blind Intubation Through The Self-Pressurised Disposable Air-Q Laryngeal Intubation Mask: An International Multicentre Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0151
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Elective Surgery Requiring Tracheal Intubation Using an Oral Tracheal Tube

ARMS (1):
- Air-Q Intubation Laryngeal Mask (Experimental): Patients will be intubated using the Air-Q Intubation Laryngeal Mask and subsequently intubated with a commercially available endotracheal tube via the Intubation Laryngeal Mask.
  Interventions: Device: Air-Q Intubation Laryngeal Mask

INTERVENTIONS:
Device: Air-Q Intubation Laryngeal Mask — Patients will be intubated using the Air-Q Laryngeal Mask.

SUMMARY:
The disposable Air-Q self-inflating laryngeal intubation mask (Air-Q, Mercury Medical, Clearwater, FL, USA) is an extra-glottic airway device which enables blind intubation with a tracheal tube. This intubating laryngeal airway device (ILA) is already commercially available and worldwide certificated (CE 0482), but data about the success rates of blind intubation via this device in adult patients are lacking. Success rates of blind intubations with the non-self-inflating device range between 57 and 97%.

Although the self-inflating disposable Air-Q device is certified for blind intubation, the success rate and rate of adverse events associated with this procedure have not been published so far. In a study comparing adverse events of conventional intubation with blind intubation via a different supra-glottic airway device (ILMA) the rates of sore throat and cough were comparable in both groups and were reported in 10-17% of the patients. In a pilot study using the non-self-inflating Air-Q for blind intubation in 19 patients, 10% reported dysphagia and one patient had a bilateral lingual nerve injury which was self-limited. One study using the self-pressurised disposable Air-Q for ventilation of children showed broncho- or laryngospasm in 3% and mucosal damage such as blood stained ILA or sore throat were reported in 1%.

This data suggests that the rate of adverse events using the Air-Q supra-glottic device are comparable to other devices such as LMA.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* elective surgery requiring tracheal intubation using an oral tracheal tube
* anticipated extubation in the operating room
* American Society of Anaesthesiologist Physical Status 1-3
* age = 18 years and = 85 years
* oral and written informed consent
* weight = 100kg (according to the product description)
* ability to understand the study information

Exclusion criteria:

* pharyngeal, laryngeal or tracheal pathology, including tracheostomy
* mouth opening < 2.5 cm
* any form of airway infection such as upper-respiratory tract infection, pneumonia or suspected tuberculosis
* any disease that might impair the power of judgement (psychiatric disease, dementia)
* indicated rapid sequence induction which is a standard when high risk for regurgitation and/or aspiration is present
* the subject must not be involved in any other clinical trial during the course of this trial, nor within a period of 30 days prior to its beginning or 30 days after its completion
* pregnancy
* breast feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Success rate of blind intubation via the disposable Air-Q self-inflating laryngeal intubation mask. | 300 seconds
  Success is defined as placement of a tracheal tube into trachea with no more than two insertion attempts.

SECONDARY OUTCOMES:
Time for insertion of the Air-Q laryngeal mask | 300 seconds
  defined as time beginning at the moment the ILA enters the mouth until the appearance of the capnography waveform
Time for insertion of the tube | 300 seconds
  defined as the time beginning at the moment of insertion of the tube through the laryngeal mask until the appearance of the capnography waveform
First attempt rate and second attempt rate | 300 seconds
Time for removal of the Air-Q ILA device after successful intubation | 500 seconds
Rate of misplacement of the ILA | 300 seconds
Rate of misplacement of the tube | 500 seconds
risk factors of insertion failures | 500 seconds
Rate of airway injuries | 5 hours
Tightness during leak test before relaxation | 300 seconds
Tightness during leak test after relaxation | 300 seconds
Maximum drop of saturation during airway management | 500 seconds
Rate of adverse events | 5 hours
  including, but not limited to suspicion of aspiration or regurgitation (gastric fluid in the ventilation tube or hypopharynx), bronchospasm, airway obstruction, coughing, dental-, tongue-, lip- pharyngeal or laryngeal trauma
Rate of necessity of alternative airway device | 500 seconds
Rate of blood stained devices after removal of the ILA | 500 seconds
Postoperative coughing after 2 hours and the next morning | 24 hours
Postoperative hoarseness after 2 hours and the next morning | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Donat R. Spahn, Prof MD, Principal Investigator — University Hospital Zurich, Institute of Anaesthesiology
Locations (3):
- Medical University Lodz, Lodz, Poland
- Switzerland (2):
  - University Hospital Zurich, Institute of Anaesthesiology, Zurich, Canton of Zurich
  - KantonsSpital Winterthur, Winterthur